CLINICAL TRIAL: NCT06239623
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of JSI-1187 Capsule in the Treatment of Advanced Solid Tumors With MAPK Signaling Pathway Mutations
Brief Title: ERK Inhibitor JSI-1187 in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JS InnoPharm, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSI-1187-101
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor; NSCLC; Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): ERK inhibitor JSI-1187
  Interventions: Drug: JSI-1187

INTERVENTIONS:
Drug: JSI-1187 — Use ERK inhibitor JSI-1187 to treat solid tumor

SUMMARY:
JSI-1187-101 phase 1 study

DETAILED DESCRIPTION:
This study is a multicenter, open-label, dose-escalation and dose- expansion phase I clinical study. To investigate the safety, tolerability and PK characteristics of JSI-1187 capsule in Chinese patients with advanced solid tumors harboring MAPK signaling pathway mutations, and to evaluate the efficacy of JSI-1187 capsule in the treatment of advanced solid tumors harboring MAPK signaling pathway mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Age of both sexes ranged from 18 to 75 years (inclusive of 18 and 75 years old).
2. For dose escalation phase only:

   Patients with locally advanced or metastatic solid tumors with histologically or cytologically confirmed MAPK signaling pathway mutations who are unresponsive to standard treatment regimens or for whom no standard treatment regimens are available;
3. Only in the extension stage (all the following conditions must be met):

   Patients who have histologically or cytologically confirmed, locally advanced or metastatic solid tumors with the following MAPK signaling pathway mutations that do not respond to or have no standard treatment options:

   Locally advanced or metastatic head and neck cancer, melanoma, small bowel cancer, bile duct cancer, and gallbladder cancer with BRAF non-V600 (G469, L597, L485, etc.) mutation (approximately 10-30 cases, subject number adjusted according to efficacy); Locally advanced or metastatic colorectal cancer, cholangiocarcinoma, gallbladder cancer, small bowel cancer or other solid tumors with BRAF V600 E mutation (approximately 10-20 cases, of which colorectal cancer is expected to be 3-6 cases, the number of subjects will be adjusted according to efficacy); KRAS G12V-mutated, locally advanced or metastatic non-small- cell lung cancer (approximately 10 patients, adjusted for the number of participants according to efficacy).
4. ECOG performance status (Appendix 2) is 0-2.
5. Life expectancy of ≥12 weeks.
6. patients should have adequate end-organ function, with laboratory results 7 days before the first dose meeting the following requirements: Bone marrow reserve: absolute neutrophil count (ANC) ≥1.5×109/L, platelet ≥100×109/L, and hemoglobin ≥90 g/L;(no use of hematopoietic stimulating factors such as EPO, G-CSF or GM-CSF in the 14 days before the test, and no blood transfusion in the 14 days before the test) Liver function: serum albumin ≥3.0 g/dL; Total bilirubin ≤1.5× upper limit of normal value (ULN), ALT and AST≤ 2×ULN, if liver metastasis or liver cancer patients, ALT or AST≤3×ULN; Renal function: creatinine ≤1.5×ULN or creatinine clearance ≥60 mL per minute (according to the Cockcroft-Gault formula; see Appendix 3); Coagulation function: INR≤1.5×ULN, APTT ≤1.5×ULN.
7. Cardiac function: left ventricular ejection fraction (LVEF)≥50%.
8. Female or male participants of childbearing age and their partners are required to use a medically approved contraceptive method (Annex 4) during the study treatment period and for 3 months after the end of the study treatment period if the women of childbearing age (defined as those younger than 50 years old or older than 50 years of age who are amenorrheic for less than 12 months before screening) tested negative for serum β-HCG.
9. Participants are required to provide informed consent for the study and to sign an informed consent form before the trial.
10. At least one measurable lesion was present according to RECIST 1.1 criteria

Exclusion Criteria:

1. Patients with a history of allergy to any component of JSI-1187 or its pharmaceutical excipients.
2. Patients with prolonged QTcF (QTcF: male >450 ms, female >470ms, QTcF formula is shown in Appendix 5).
3. Patients who has previously received other ERK inhibitors.
4. Active central nervous system tumors or central nervous system metastases, as indicated by clinical symptoms, cerebral edema, need for systemic hormone use, and disease progression. Patients with treated tumors or metastases of the central nervous system are eligible if they have been clinically stable (as determined by imaging or other clinical testing) for at least 8 weeks and if they had stopped immune suppressive systemic hormones (> 10 mg per day of prednisone or equivalent) for at least 4 weeks before the first dose of study drug.
5. Patients with basal-cell, squamous-cell, or carcinoma in situ are excluded if they had a history of other malignancies within 2 years before enrollment, have undergone potentially curative treatment, and have been free of disease recurrence for 5 years after the initiation of treatment.
6. History of or current evidence/risk of retinal vein occlusion or central serous retinopathy.
7. Have received antineoplastic therapy within 28 days before the first dose, including but not limited to: chemotherapy, biotherapy, radiotherapy (except palliative radiotherapy for patients with bone metastases), endocrine therapy, targeted antineoplastic therapy (except nitrosourea and mitomycin C); Received nitrosourea or mitomycin C within 6 weeks before the first dose. Had received treatment with a traditional Chinese medicine with definite antitumor effects within 14 days before the first dose. Except for alopecia and eligibility criteria, radiation-related toxicities (including radiodermatitis dermatitis, post-radiation recall reactive dermatitis, soft tissue fibrosis, etc.) did not recover to grade 1 or lower (according to CTCAE 5.0) after palliative radiotherapy in patients with bone metastases.
8. Patients have received other drugs which are still in clinical trials within 28 days before the first dose.
9. Patients who has undergone major surgical procedures or has active ulcers (which are still present) or wounds that do not fully heal within 28 days before the first dose.
10. Chronic systemic comorbidities (e.g., severe chronic lung, liver, kidney, or heart disease) that cannot be controlled (have received active treatment but is not currently stable or may progress/relapse during the trial).
11. Patients with severe cardiac disease, such as uncontrolled arrhythmia, myocardial infarction, unstable angina, or New York Heart Association (NYHA) class III-IV cardiac dysfunction, within 6 months prior to the first dose (Annex 6).
12. Patients who have factors that increase the risk of QTc prolongation and the risk of arrhythmias, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, sudden death of an immediate family member under 40 years of age from an unknown cause, and taking any concomitant medications that cause prolongation of the QT interval (Appendix 7).
13. Patients with uncontrolled (actively treated but not currently stable or with potential disease progression/recurrence during the trial) body fluid (pleural effusion, pericardial effusion, or ascites).
14. Patients who are in the acute phase of infection and require medical therapy.
15. Unable to swallow capsules or suffering from a condition that significantly affects gastrointestinal function, such as malabsorption syndrome, gastric or small bowel resection, symptomatic inflammatory bowel disease, partial or complete bowel obstruction.
16. Patients who are taking (or could not be discontinued 2 weeks before the first dose) any known strong inhibitor or strong inducer of CYP3A4, BCRP substrate, or who needed to continue receiving these drugs during the study (Appendix 8).
17. Positive human immunodeficiency virus antibody (HIV-Ab) within 1 week before the first dose; Or HCV antibody (HCV-Ab) positive and HCV RNA quantification > the upper limit of normal value of the detection unit;Or patients with positive hepatitis B surface antigen (HBsAg) and HBV DNA > the upper limit of normal value.
18. The presence of serious psychological or psychiatric abnormalities that affect the patient's compliance to participate in this clinical study.
19. Patients with a history of psychotropic substance abuse or drug use.
20. Patients with adverse event worse than CTCAE1 that is not resolved due to previous antineoplastic therapy before the first dose (except alopecia, sensory neuropathy, and eligibility criteria otherwise required).
21. Women who are lactating.
22. Any other condition judged by the investigator to be inappropriate for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2024-09-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | through study completion, an average of 1 year
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.
Serious Adverse Events | through study completion, an average of 1 year
  Any untoward medical occurrence that at any dose:results in death、is life-threatening、requires inpatient hospitalization or prolongation of existing hospitalization、results in persistent or significant disability/incapacity,or is a congenital anomaly/birth defect

SECONDARY OUTCOMES:
Objective Response Rate | through study completion, an average of 1 year
  The proportion of patients with complete and partial responses.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PhD, Principal Investigator — Beijing Cancer Hosptial
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China